CLINICAL TRIAL: NCT02129335
Title: Stress, Exercise Behavior and Survival in Patients With Newly Diagnosed Glioblastoma and in a Close Partner (TOGETHER-study): a Prospective Multicenter Cohort Study.
Brief Title: Stress, Exercise Behavior and Survival in Patients With Newly Diagnosed Glioblastoma and in a Close Partner
Acronym: TOGETHER
Status: Terminated | Type: Observational
Why Stopped: insufficient enrollment
Sponsor: University Hospital, Basel, Switzerland (Other)
Collaborators: University Hospital, Zürich (Other); Luzerner Kantonsspital (Other); Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Sponsor
Other Study IDs: TOGETHER
Record Dates: First submitted 2014-04-07; First posted 2014-05-02 (Estimated); Last update posted 2017-05-17 (Actual); Status verified 2017-05

CONDITIONS: Neoplasms; Glioblastoma
Keywords: glioblastoma; partner; stress; exercise; outcome
MeSH Terms: conditions — Neoplasms; Glioblastoma; Motor Activity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- stress: patient with glioblastoma diagnosis and partners
  Interventions: Other: stress

INTERVENTIONS:
Other: stress — stress level and survival

SUMMARY:
Glioblastoma multiforme (GBM) is the most common malignant central nervous system (CNS) tumor in adulthood with a median survival of 12-16 months. The drastically shorted life expectancy, intellectual changes and rapid physical decline in those patients are devastating and do impose a profound chronic stress on patients and their families. There is extensive evidence that chronic stress can promote cancer growth and progression. In the setting of GBM patients, three major questions still have to be answered and will be analysed in this study:

1. Is there a prognostic significance of stress in patients with newly diagnosed GBM on treatment tolerance and (progression free) survival?
2. Can this stress be modulated by other factors, like stress of patients partners and patients physical activity, a known independent prognostic factor in recurrent glioma patients?
3. How is the longitudinal course of patients and partners stress and physical condition over the disease course and do they influence (progression free) survival?

Answers to these questions will help to establish future projects studying non drug interventions in patients and patients partners to help improving clinical and tumor related outcome in patients with newly diagnosed GBM.

The investigators hypothesize that chronic stress, specifically measured as a disruption of the diurnal cortisol rhythmicity, is an independent prognostic factor in patients with GBM. Furthermore, physical activity of patients and stress level in patients' partners may impact - as stress-modulating factors- on stress in patients and on their prognosis.

Aiming at identifying stress-related prognostic factors as potential targets for novel treatment approaches, we propose, in a first step, a prospective multicenter cohort study: all patients with newly diagnosed GBM and good performance status (KPS ≥ 50%) who undergo standard treatment with combined radiochemotherapy with temozolomide (RCT) followed by 6 month of cyclic temozolomide, are eligible. In addition, one "partner", defined as a close person living in the same home or close daily contact to the patient, will be asked for inclusion.

DETAILED DESCRIPTION:
General Aim The aim of this prospective, multicenter observational cohort study is to determine the impact of baseline bio-behavioral stress (Aim I) on cancer progression and survival in patients with newly diagnosed glioblastoma (GBM) undergoing standard radiochemotherapy. The role of baseline physical activity (PA) and baseline partner's distress as stress-modulating factors will be assessed in an exploratory analysis.

Secondary aims include a longitudinal assessment of self-reported psychological distress in this homogenous patient cohort and their partners (Aim II) and -in a translational subproject - to determine the role of serum copeptin as a biomarker for distress (Aim III).

Specific Aims Specific Aim I: Prognostic role of stress at the time of diagnosis in GBM patients In this analysis, baseline neuroendocrine stress will be correlated to progression-free survival (PFS).

More specifically we aim at assessing

IA) Whether stress-induced disruption of diurnal cortisol rhythmicity as measured by the salivary cortisol slope is an independent prognostic factor for (progression-free) survival in patients with newly diagnosed GBM undergoing standard multimodal treatment.

IB) Whether increased baseline self-reported physical activity is correlated with lower levels of stress (i.e. acts as a stress-modulating factor) and prolonged (progression-free) survival

IC) Whether high levels of stress in the patients' partner (baseline diurnal cortisol slope) are correlated with high levels of stress in the patient (i.e. stress-modulating factor) and shorter (progression-free) survival

Specific Aim II: Longitudinal cohort of patient-partner dyads In the same cohort of patients (Aim I above) we aim at describing distress over time (three-monthly) from start of combined radiochemotherapy to disease progression in patients and - as a paired dyad - in one close partner.

Specific Aim III: Copeptin biomarker subproject In a translational subproject we aim at assessing the prognostic role of baseline serum copeptin- an easy to test serum biomarker of stress in many clinical situations, which has never been assessed in cancer patients.

Methods Study design Since the prognostic role of stress in GBM has not been studied before, we propose in a first step an observational, prospective multicenter cohort study in a well-defined group of patients, all at the same stage of disease (initial diagnosis) and all undergoing the same standard multimodal treatment (surgery followed by radiochemotherapy according to R.Stupp et al.).

Patients All patients in good performance status (Karnofsky Performance Score (KPS) ≥ 50%), aged 18 years and older, with histologically confirmed, previously untreated GBM are eligible prior to starting initial treatment with radio-chemotherapy. In order to participate, patients will need to have given their informed consent on the ethics-approved consent form and will need to be willing and able (as judged by the investigator) to comply with the protocol. Cardiovascular contraindications to the 6-minute walking test (6MWT) and/or a history of instable angina pectoris or New York Heart Association (NYHA) grade II or greater congestive heart failure (according to the Thoracic Society recommendations) preclude trial inclusion. Equally, patients who have signs or symptoms (including laboratory findings) of conditions, either metabolic or psychological, that interfere with adequate assessment of the stress axis (e.g. chronic use of a corticosteroid, psychiatric disorder and medication) are excluded. Perioperative dexamethasone treatment is not an exclusion criterion as short time treatment does not clearly affect the HPA axis and synthetic corticosteroids can be discriminated in salivary cortisol measurements. Inability to follow study procedures, e.g. due to language problems, psychological disorders, dementia or confusion, is another reason for study exclusion.

Patients' partners Each patient designates his or her closest partner, (not necessarily intimate partners), either a person living in the same household or with daily contact (husband/wife, not married partner, other family members). In order to participate, the patient's partner must be older than 18 years, in a good performance status (KPS≥50%), willing and able (as judged by the investigator) to comply with the protocol and must give informed consent.

If the patient has no partner or the partner is not willing to be part of the trial, participation in the cohort is still possible (the group of patients without partners will be analyzed separately).

Primary Endpoint for Aim I The primary endpoint is PFS, i.e. the time between diagnosis and disease progression (according to RANO criteria) or death of any cause.

Response evaluation in MRI will be done using the criteria by MacDonald et al. , which are specified in the RANO criteria. In brief, the definitions for "progression" is the following: At least 25% increase in the size of a solid mass or contrast-enhancing lesions on MRI (or CT) or the appearance of a new lesion or clinical deterioration.

Secondary Endpoints for Aim I

Secondary endpoints include overall survival and measures of treatment tolerance:

* Number of patients, who stopped treatment for reasons other than progressive disease
* Percentage of planned temozolomide doses received

Study Flow and Assessments

Assessments Baseline (T1): predictor variables Baseline Assessment will occur at a strictly defined time point (T1) in order to minimize time-dependent confounders on predictor variables (particularly stress lab): Physical functioning tests and questionnaires will be performed on days -3 before start of radiochemotherapy. Salivary cortisol samples will be performed at days -2 and -1 before start of radiochemotherapy.

Baseline Consolidation (T2) The visit will take place 28d after T1 when patients have started their treatment ("steady-state"), for all non-progressing patients (which will be the vast majority at this early time-point) and includes the same assessments as T1. The purpose of T2 assessments is to validate T1 i.e. to confirm that T1 (baseline) has been representative for the condition patients and partners are in early during treatment and to exclude that T1 assessments have been unrepresentative due to the impending start of an unknown treatment. T2 assessments will be analyzed as confirmatory baseline prognostic factors in all non-progressing patients.

Follow up visits until progression (FU1) Follow-up visits will be done every 12 weeks. The purpose of the FU1 visits is i) to measure disease status in MRI for aim I (1° endpoint) and ii) to longitudinally describe distress, emotional functioning and quality of life (QoL) in patients and partners for aim II.

Follow up visits from progression to death (patients only) (FU2) After progression patients will be contacted every three months for survival status (dead or alive).

Study procedures Stress Aim I (predictor variables): Baseline Stress measurements in patients as well as partners at baseline (T1) and after 4 weeks (T2) i) Neuroendocrine stress evaluations using standard laboratory essays (salivary diurnal cortisol slope, cortisol awakening response (CAR), short adrenocorticotropic hormone (ACTH)-test as well as ii) Self-reported psychological distress evaluations by questionnaires (distress thermometer and perceived stress scale)

Aim II (descriptive variables): Distress in the longitudinal cohort will be evaluated every three months in patients-partners dyads with self-reported measures such as DT and PSS (ii above). Quality of life and emotional functioning will also be described as measured by the FACT-Br and HADS-D score

Ad i.)

* Diurnal Cortisol Slope: Salivary cortisol levels peak 30-60 minutes after awakening and then drop to a nadir during sleep. This diurnal rhythm is disrupted in chronically stressed patients: leading to a flattening of the slope (beta) of the curve that connects salivary cortisol concentrations over time (from awakening to bedtime). Salivary cortisol will be measured on two consecutive days (patients will receive a kit with "salivettes" containers to use at home and store in the refrigerator until next day hospital visit). Salivary samples will be collected after waking up in the morning, 30 minutes later (for CAR below), at 4pm and at 9pm. Cortisol level analyses will be done by the immunoassay ECLIA (E170 Roche, Switzerland) at the reference hospital (University Hospital Basel). Sample storage and shipment can be performed at -20°C.
* The cortisol awakening response (CAR) describes the increase of about 50% in saliva cortisol levels, which occurs 20-30 minutes after waking up in the morning. It is thought to be linked to the hippocampus' preparation of the hypothalamic-pituitary-adrenal axis (HPA) to face anticipated stress and it is independent from the circadian variation in the HPA axis. CAR provides an easy measure of the capacity of the HPA axis to react to stress. An increased CAR has been associated with burnout, worry and chronic stress at work. For CAR saliva samples will be collected on two consecutive days by passive drooling, immediately after awakening (0') and 30 min (30') later [45].
* As perioperative dexamethasone is usually given in these patients, a short or "low-dose" ACTH test (Synacthen test) will be performed, to rule out relative adrenal insufficiency. The test reflects the adrenal function and is a validated and save tool routinely used in daily practice. A baseline sampling of Cortisol is performed before 1 ug Synacthen is applied by intravenous route. Stimulated Cortisol serum level is measured exactly 30min after Synacthen application. The test will be performed in the morning. Cortisol level analyses will be done by the immunoassay ECLIA (E170 Roche, Switzerland).

Ad ii) The distress-thermometer (DT) is a 10-point scale displayed in a thermometer format and was originally developed by Roth and colleagues (Appendix 1). Validity of DT has been examined for outpatient cancer patients as well as relatives.

The perceived stress scale (PSS) is a universally accepted, standardized unidimensional scale that assesses perceived stress by asking respondents to report whether their lives seem to be unpredictable or uncontrollable, or if they feel overburdened. It assesses the cognitively mediated emotional response to an objective event, rather than the objective event itself.

Quality of life (QOL) will be measured with the Functional Assessment of Cancer Therapy (FACT). The FACT comprises a series of questionnaires to measure general QOL, as well as cancer- and condition-specific symptoms during and after cancer treatment. The questionnaires are broadly used and validated in several languages, including German. The following scales will be used: FACT-Br (brain), containing 37 items on physical wellbeing, family/social wellbeing, emotional wellbeing and functional wellbeing. For comparable evaluations in partners, an adapted version of the FACT-G (general) has been generated.

Emotional functioning: The German version of the Hospital Anxiety and Depression Scale (HADS-D) will be used to assess current levels of depression and anxiety. Each scale comprises 7 items, which are answered on a 4-point scale. The scale is widely used to evaluate emotional wellbeing in patients with chronic physical conditions and is validated for the German language.

Physical activity Exercise behavior will be evaluated in patients as well as in partners by self-reported physical activity in MET-hours per week, by Godin-Leisure-Time-Exercise Questionnaire (GLTEQ). In this questionnaire -validated in glioma patients- patients and partners are asked to complete a self-explanatory four-item query of usual leisure-time exercise habits.

-Physical condition (in patients only) will be tested using an internationally standardized test that does not need extensive equipment (which is important for practicability in the multicenter setting): A 6-Minute walking test (6MWT) is a simple method to evaluate functional capacity and has been tested in multiple settings. Patients will be instructed to walk at their fastest pace and to cover the longest possible distance over 6 minutes under the supervision of physical therapist. During exercise, oxyhemoglobin saturation and heart rate will be monitored by pulse oximetry.

Aim III: Copeptin Arginine Vasopressin (AVP) is a hypothalamic stress hormone, which is produced in the hypothalamus and released from the posterior pituitary. Together with corticotropin-releasing hormone, it leads to secretion of ACTH and cortisol. With the recent development of a novel sandwich immunoassay for copeptin (the C-terminal glycoprotein of the pre-provasopressin), a stable and easy to measure surrogate of AVP secretion has become available. (Direct AVP measurement is hampered by technical, pre-analytical difficulties). As a stress hormone copeptin mirrors individual stress levels even more subtly than cortisol.

ELIGIBILITY:
Inclusion Criteria:

Patients:

* age ≥18 years
* Karnofsky Performance Score ≥ 50 %
* histologically confirmed, previously untreated GBM
* radiochemotherapy according to Stupp et al [1] is planned (ideally, treatment start can be scheduled on a Monday)
* no cardiovascular or neurological contraindications for 6MWT and/or a history of instable angina pectoris or NYHA grade II or greater congestive heart failure (according to the Thoracic Society recommendations [2])
* willing and able to comply with the protocol as judged by the investigator
* signed informed consent

Partners:

* age ≥18 years
* willing and able to comply with the protocol as judged by the investigator
* spouse or partner living in the same home as the patient or closest contact as named by the patient (1-2h 5 days a week)
* signed informed consent

Exclusion Criteria:

Patients:

* Patients who have any other disease, either metabolic or psychological, or who have any evidence on clinical examination or special investigations (including laboratory findings) which give reasonable suspicion of a condition that interferes with the adequate measurement of the stress axis (e.g. chronic use of corticosteroids ≥ 3 months before study entry for disease other than glioblastoma, (dexamethasone use in the context of glioblastoma is allowed)
* Severe, medically treated psychiatric disorder prior to the diagnosis of glioblastoma
* Participation in a study with investigational drugs
* Severe asthma or known allergy against tetracosactide (Synacthen®)
* Pregnancy or breast feeding
* Inability to follow the procedures of the study, e.g. due to language problems, psychological disorders, neurologic deficits that interfere with the planned walking tests, dementia or confusional state

Partners:

* Individuals who have any disease, either metabolic or psychological, that interferes with the adequate measurement of the stress axis (e.g. chronic use of corticosteroids (≥ 3 months), psychiatric disorders)
* Pregnancy or breast feeding
* Inability to follow the procedures of the study, e.g. due to language problems, psychological disorders, dementia or confusional state

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Newly diagnosed GBM with one Partner.
Sampling Method: Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2014-04; Primary Completion 2016-10 (Actual); Study Completion 2017-05 (Actual)

PRIMARY OUTCOMES:
Progression free survival | 12 month
  analysis

SECONDARY OUTCOMES:
Overall survival | 12 month
  analysis

CONTACTS AND LOCATIONS:
Overall Officials: Viviane Hess, MD, Study Chair — University Hospital, Basel, Switzerland; Katrin Conen, MD, Principal Investigator — University Hospital, Basel, Switzerland
Locations (3):
- Switzerland (3):
  - University Hospital Basel, Basel
  - Kantonsspital Luzern, Lucerne
  - University Hospital Neurology, Zurich